CLINICAL TRIAL: NCT00864110
Title: A Multi-Center Phase 1b Pharmacokinetic and Radiation Dosimetry Study Evaluating 99mTc-EC-DG SPECT/CT in Patients With Non-small Cell Lung Cancer (NSCLC)
Brief Title: Pharmacokinetic and Radiation Dosimetry Study Evaluating 99m TC-EC-DG SPECT/CT in Patients With Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cell>Point LLC (Industry)
Collaborators: Numoda (Industry); Venn Life Sciences (Other); Camargo Pharmaceutical Services (Industry); Biomedical Systems (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CP-05-233
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non small cell lung cancer; SPECT CT imaging; Pharmacokinetic; Radiation Dosimetry; PET CT comparison
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — technetium 99m ethylenedicysteine deoxyglucose; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 99mTc EC-DG (Experimental): 99mTc-EC-DG with SPECT/CT imaging
  Interventions: Radiation: Radiolabeled (99Tc) EC-DG (ethylenedicysteine-deoxyglucose); Radiation: Technetium 99m ethylenedicysteine-deoxyglucose
- 18F FDG (Active Comparator): 18F FDG with PET/CT imaging
  Interventions: Radiation: 18 F fluorodeoxyglucose

INTERVENTIONS:
Radiation: Radiolabeled (99Tc) EC-DG (ethylenedicysteine-deoxyglucose) — one injection of Technetium ethylenedicysteine-deoxyglucose to yield a target activity of 20 mCi (range 20-30 mCi) to be given by slow IV push (over 3-5 minutes) 1mg of EC-DG will be injected
  Arms: 99mTc EC-DG
Radiation: Technetium 99m ethylenedicysteine-deoxyglucose — 99mTc EC-DG injection, single dose, slow IV push over 3-5 minutes, yielding a target activity of 20 mCi (range 20-30 mCi)
  Arms: 99mTc EC-DG
Radiation: 18 F fluorodeoxyglucose — single injection of 18F FDG (range 10-20 mCi)
  Arms: 18F FDG

SUMMARY:
This is a multi-center Phase 1 b study designed to expand the patient safety using 99mTc-EC-DG with SPECT/CT imaging and to expand the patient radiation dosimetry and pharmacokinetic database using 99mTc-EC-DG in patients who have non-incisional biopsy definitive evidence of Non-small Cell Lung Cancer as compared to 18F-FDG PET/CT imaging.

DETAILED DESCRIPTION:
Male and female patients at least 18 years old with untreated Non-small Cell Lung Cancer who have non-incisional biopsy definitive evidence of disease (or cytology results from a bronchoscope procedure confirming NSCLC) and who have been previously certified (per Centers for Medicare and Medicaid Services requirements)by their physicians will be consented for the study. The study consists of a screening visit, gold-standard 18F-FDG PET/CT imaging followed by the investigational agent 99mTc-EC-DG with SPECT/CT(if the PET/CT was performed as part of the pre-study activities on a qualified PET camera for this study, the SPECT/CT must be done within 45 days of the PET/CT imaging procedures). The study procedures can be performed within 5-7 days of signing the informed consent. During the 99mTc-EC-DG SPECT/CT visit of the study, pharmacokinetic (PK) blood draws and urine collection will be taken and radiation dosimetry (Planar Imaging) will be performed at specified time points post 99mTc-EC-DG injection. Patients will be seen 24 hours after the 99mTc-EC-DG injection for safety and final PK blood and urine collection. A 21-day follow-up period (after the SPECT/CT image) will allow the investigator to acquire additional imaging, surgical, pathology and treatment documentation (an actual patient visit is not required at the 21 day follow-up time point).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients at least 18 years old;
* Have non-incisional biopsy demonstrating definitive evidence for NSCLC and have not been treated for lung cancer (surgery, radiation and/or chemotherapy). A copy of the actual report must be requested by the patient through a medical release form if not already done. The copy must be available to the study doctor within 28 days of the screening visit/ Visit 1 ;
* Be certified as per Centers for Medicare and Medicaid Services (CMS) requirements and be eligible for a PET scan;
* Have an Eastern Co-operative Oncology Group (ECOG) performance rating ≤ 2 (see Appendix 1);
* Males or non-pregnant, non-lactating females who are postmenopausal, naturally or surgically sterile, or who agree to use effective contraceptive methods throughout the course of the study. Postmenopausal is defined as at least 12 months natural spontaneous amenorrhea, or at least 6 weeks following surgical menopause (bilateral oophorectomy);
* Females of childbearing potential and males with female sexual partners of childbearing potential must agree to use one of the following acceptable birth control methods:

  1. Surgically sterile (hysterectomy or bilateral oophorectomy);
  2. Surgically sterile (bilateral tubal ligation with surgery at least 6 weeks prior to study initiation). Documentation is required;
  3. Intrauterine device (IUD) in place for at least 3 months;
  4. Double-barrier method (condom and diaphragm) with spermicide for at least 14 days prior to screening and through study completion;
  5. Stable hormonal contraceptive (oral, topical, vaginal or implanted/injected) for at least 3 months prior to study and through study completion;
  6. Abstinence;
  7. Single-barrier method for at least 14 days prior to screening and though study completion for vasectomized males or females with vasectomized partners;
* Have a fasting blood glucose of less than 200 mg/dL at screening;
* Have reported clinical symptoms consistent with a confirmed diagnosis of NSCLC;
* Be able to tolerate SPECT/CT and PET/CT imaging. This includes:
* Laying in the same position without moving for approximately 45 minutes;
* Able to tolerate a claustrophobic area;
* Ability to hold their arms overhead for approximately 45 minutes;
* Be able to fast prior to SPECT/CT and PET/CT imaging, with length of fasting dependent on the time of the scan:

  * A morning scan (08:00-12:00) will require fasting from midnight (or as per the site's fasting/diet restrictions);
  * An afternoon scan (12:00-onward) will require a minimum 6 hour fast (or as per the site's fasting/diet restrictions);
* Be able to eat a high protein/low carbohydrate meal as the last meal before SPECT/CT and PET/CT imaging (or as per the site's fasting/diet restrictions);
* Be able to make the scheduled appointments within the designated time windows [PET/CT imaging within 7 days of qualifying for the study, the second imaging session with SPECT/CT imaging 1 - 3 days after the initial imaging visit, with at least 24 hours between PET/CT and SPECT/CT imaging (if the PET/CT is performed as part of pre-study activities on a qualified PET camera for this study, the SPECT/CT must be done within 45 days of the PET/CT imaging procedure)];
* Have safety laboratory values that in the opinion of the Investigator do not place the patient at undue risk if the patient were to participate in the study. This includes (but is not limited to):

  * Alanine aminotransferase 2.5 × upper limit of normal (ULN);
  * Aspartate aminotransferase 2.5 × ULN;
  * Creatinine 2.5 × ULN;
  * Bilirubin 2.0 × ULN;
* Able to understand and provide signed informed consent;
* Females of childbearing potential must have a negative urine or serum β-human chorionic gonadotropin (hCG) pregnancy test at screening.

Exclusion Criteria

* Any clinically significant safety concerns (laboratory, electrocardiogram [EKG], physical examination, other) that, in the opinion of the Investigator, would place the patient at undue risk if the patient were to participate in the study;
* Undergoing any current treatment for cancer (radiation therapy, surgery or chemotherapy)
* Diabetic with insulin dependence (Patients who have a known insulin dependence for diabetes can be included in the study if the standard of care protocol in place at the clinical site provides for the management of the patient's glucose level sufficiently to allow the PET/CT imaging to be performed. The same glucose management used for the PET/CT imaging should be applied to the SPECT/CT imaging procedures. A waiver will be required to be completed by the clinical site and approved by the sponsor or designee);
* Patient weight above the SPECT/CT and PET/CT table weight limit;
* Failure to have a non-incisional biopsy definitive diagnosis (or cytology report from a bronchoscope) for NSCLC (a copy of the biopsy/cytology report must be available to the investigator within 28 days of Visit 1);
* Will not agree to use an effective means of contraception for the duration of the study (males and females);
* Known hypersensitivity to EC-DG or FDG or similar compounds including any of the inactive ingredients;
* Known or suspected pregnancy, lactation or planned pregnancy (females and male partners);
* Clinically significant mental illness (to be determined by the Investigator);
* Exposure to any investigational agent within 30 days prior to screening visit or participating in an ongoing clinical study (this criteria can be overruled by the Principal Investigator with appropriate documentation of the reason for the exception);
* Patient has a condition the Investigator believes would interfere with the ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results or put the patient at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Safety: through adverse event collection | from 99mTc-EC-DG injection through 21 days

SECONDARY OUTCOMES:
Pharmacokinetic (blood) | 0 hour, post-injection:15 minutes, 1, 2, 4, 6, 24 hours
Pharmacokinetic (urine) | pre-injection, 0-2, 2-4, 4-6, 6-24 hours post injection
Radiation Dosimetry (whole body planar imaging) | 15 minutes, 2, 4, 6 hours post injection
Comparison of the results of EC-DG:SPECT/CT (als) to biopsy results and FDG:PET/CT (als) | At end of study

CONTACTS AND LOCATIONS:
Overall Officials: Donald Blaufox, MD, Principal Investigator — Albert Einstein University, Montefiore Medical Center
Locations (3):
- United States (3):
  - University of Chicago, Chicago, Illinois
  - Mayo Clinic, Division of Nuclear Medicine, Rochester, Minnesota
  - Montefiore Medical Center, The Bronx, New York

REFERENCES:
- See also: Location of the study — http://mayoclinic.com
- See also: Sponsor link — http://cellpointweb.com